CLINICAL TRIAL: NCT01662310
Title: Paliperidone Extended Release Tablets for the Prevention of Relapse in Subjects With Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study
Brief Title: An Efficacy Study of Paliperidone for the Prevention of Relapse in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100427; R076477-SCH-3041 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-03-29; First posted 2012-08-10 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Paliperidone Extended-Release
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paliperidone: Run-in or Stabilization phase (Experimental): Paliperidone extended-release (ER) oral tablet will be administered at a starting dose of 3 milligram (mg) once daily for 8 weeks. Dose will be increased from milligram per day (3 mg/day) after 5 days based on Investigator's discretion, up to maximum of 12 mg/day.
  Interventions: Drug: Paliperidone
- Paliperidone: Double blind (DB) phase (Experimental): Participants who transitioned from run-in or stabilization phase received 3 to 12 mg fixed dose of paliperidone ER oral tablet once daily during DB phase of the study. Participants who will experience a relapse event during the DB phase or who will remain relapse free for the entire duration of the DB phase and participants, who will be enrolled at the time the study termination will enter in open label extension phase, wherein paliperidone ER oral tablet will be administered once daily as 3 to 12 mg.
  Interventions: Drug: Paliperidone
- Placebo: DB phase (Active Comparator): Participants who transitioned from run-in or stabilization phase received matching placebo to paliperidone ER once daily during DB phase of the study. Participants who will experience a relapse event during the DB phase or who will remain relapse free for the entire duration of the DB phase and participants, who will be enrolled at the time the study termination will enter in open label extension phase, wherein paliperidone ER oral tablet will be administered once daily as 3 to 12 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone — Paliperidone extended-release (ER) oral tablet will be administered at a starting dose of 3 milligram (mg) up to 12 mg once daily for 8 weeks in Run-in or Stabilization phase, and 3-12 mg fixed dose oral tablet will be administered in DB phase. Participants who will enter open-label extension phase will receive paliperidone as 3-12 mg per day.
  Other Names: R076477
  Arms: Paliperidone: Double blind (DB) phase; Paliperidone: Run-in or Stabilization phase
Drug: Placebo — Participants who transitioned from run-in or stabilization phase will receive matching placebo to paliperidone ER once daily during DB phase of the study.
  Arms: Placebo: DB phase

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and safety of paliperidone extended release (ER) tablets (between 3 to 12 milligram (mg), once a day) in the prevention of relapse in schizophrenia participants.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the name of the assigned drug), randomized (participants are assigned to treatment by a chance), placebo-controlled, and parallel-group study of paliperidone ER tablets. The study will consist of 6 phases: 14 days of screening phase, 8 weeks of open-label run-in phase (participants will be flexibly dosed with paliperidone ER once daily in a dose range of 3 mg to 12 mg), 6 weeks of stabilization phase (participants will continue to receive the fixed dose of paliperidone ER), double-blind (DB) phase of various length (participants will be randomly assigned in a 1:1 ratio to receive either paliperidone ER or placebo and this phase will be completed after 86 relapse events are observed or if the study is positive at the interim analysis), 6 months of open-label extension (participants who experience a relapse event or who remain relapse free for the entire duration of the double-blind phase and participants who are enrolled at the time the study is terminated, will be eligible for this phase. All participants will be treated with paliperidone ER and safety and tolerability information will be collected during this phase) phase and 6 months of follow-up phase (participants who withdraw during the DB phase for any reason other than relapse will be followed for 6 months or until they experience a relapse). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV)
* Have experienced an acute episode, with a Positive and Negative Syndrome Scale (PANSS) total score between 70 and 120 inclusive, at Screening and Baseline
* Women must be postmenopausal (for at least 1 year), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), practicing a highly effective method of birth control, if sexually active
* Men must be using a highly effective method of birth control and must not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Be willing and capable to complete the questionnaires and able to take oral medications independently

Exclusion Criteria:

* Has drug dependence diagnosis according to DSM-IV (excluding nicotine and caffeine dependence) within 6 months before screening
* Participants with Crohn's disease and hepatic or renal diseases
* Has had relevant history of any significant and/or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular dysfunction), renal, hepatic, endocrine, or immunologic diseases
* Has had history of neuroleptic malignant syndrome (the disorder caused by antipsychotic drugs with symptoms of fever, muscle rigidity and delirium)
* Has had known or suspected Stevens Johnson Syndrome (an immune disease with symptoms of fever, sore throat, ulcers and conjunctivitis) after exposure to phenytoin, carbamazepine, barbiturates, or lamotrigine
* Had been treated with clozapine for treatment refractory or treatment resistant schizophrenia
* Has significant risk of suicide or homicidal behavior, or significant risk of deliberate self harm or harm to others
* Has taken isocarboxazid, phenelzine, selegiline and tranylcypromine within 4 weeks before screening
* Has received electroconvulsive therapy within 60 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- China (14):
  - Baoding
  - Beijing
  - Changsha
  - Chengdu
  - Guangzhou
  - Harbin
  - Kunming
  - Nanjing
  - Shanghai
  - Taiyuan
  - Tianjin
  - Wuhan
  - Xi'an
  - Xinxiang

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Run-in or Stabilization Phase: Paliperidone extended-release (ER) oral tablet was administered at a starting dose of 3 milligram (mg) once daily for 8 weeks. Dose was increased from 3 milligram per day (mg/day) after 5 days based on Investigator's discretion, up to maximum of 12 mg/day.
- Paliperidone: Double Blind (DB) Phase: Participants who transitioned from run-in or stabilization phase received paliperidone at a starting dose of 3 mg up to 12 mg, fixed dose of paliperidone ER oral tablet once daily during DB phase of the study.
- Placebo: DB Phase: Participants who transitioned from run-in or stabilization phase received matching placebo once daily during DB phase of the study.
- Paliperidone DB/Paliperidone Open-label (OL) Extension Phase: Participants who transitioned from paliperidone treatment group in DB phase (that is participants who experienced a relapse event during the DB phase or who remained relapse free for the entire duration of the double-blind phase and participants, who were enrolled at the time the study was terminated), entered open label extension phase, wherein paliperidone ER oral tablet was administered once daily as 3 to 12 mg.
- Placebo DB/Paliperidone OL Extension Phase: Participants who transitioned from placebo treatment group in DB phase (that is participants who experienced a relapse event during the DB phase or who remained relapse free for the entire duration of the double-blind phase and participants, who were enrolled at the time the study was terminated), entered open label extension phase, wherein paliperidone ER oral tablet was administered once daily as 3 to 12 mg.
Period: Run-In or Stabilization Phase
Arm/Group | Paliperidone: Run-in or Stabilization Phase | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Started | 201 | 0 | 0 | 0 | 0
Completed | 136 | 0 | 0 | 0 | 0
Not Completed | 65 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 15 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Paliperidone: Run-in or Stabilization Phase | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Started | 0 | 65 | 71 | 0 | 0
Treated | 0 | 64 | 71 | 0 | 0
Completed | 0 | 50 | 66 | 0 | 0
Not Completed | 0 | 15 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 9 | 3 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Randomized but not treated | 0 | 1 | 0 | 0 | 0
Period: Open-Label Extension Phase
Arm/Group | Paliperidone: Run-in or Stabilization Phase | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Started | 0 | 0 | 0 | 47 | 59
Completed | 0 | 0 | 0 | 36 | 49
Not Completed | 0 | 0 | 0 | 11 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All the participants who were enrolled.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 91

OUTCOME MEASURES:

1. Primary Outcome: Double Blind (DB) Phase: Median Time to Relapse
Description: A relapse is defined as any one of the following: 1. involuntary or voluntary psychiatric hospitalization 2. deliberate self-injury or violent behavior; 3. Suicidal or homicidal ideation and clinically significant aggressive behavior; 4. 25 percent (%) increase in Positive and Negative Syndrome Scale (PANSS) total score for 2 consecutive assessments for participants whose score was greater than 40 at randomization, or a 10-point increase for participants who scored less than or equal to (≤) 40 at randomization; 5. increase for 2 consecutive assessments in PANSS items (delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, hostility or uncooperativeness) to greater than or equal to (≥) 5 for participants who scored ≤3 at randomization, or to ≥6 for participants with initial score of 4. Independent Data Monitoring Committee performed ongoing safety monitoring during double-blind treatment and conducted the interim analysis after 61 relapse events had taken place.
Time Frame: DB Baseline (Day 1 of Week 15) up to interim analysis data cut-off (24 August 2012) (Approximately 1 year)
Population: The Intent-to-Treat DB analysis set included all the participants who were randomized into the DB phase and who received at least one dose of DB study medication up to interim analysis cut-off date (24-Aug-2012). "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Paliperidone: Double Blind (DB) Phase: Participants who transitioned from run-in or stabilization phase received 3 to 12 mg fixed dose of paliperidone ER oral tablet once daily during DB phase of the study.
- Placebo: DB Phase: Participants who transitioned from run-in or stabilization phase received matching placebo to paliperidone ER once daily during DB phase of the study.
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 59 | 65
Days | NA [NA to NA] — Median time was not reached as data was not matured at the time of the analysis, hence no data could be reported. | 49.0 [22.0 to 77.0]

2. Secondary Outcome: Run-In and Stabilization Phase: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 14
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Week 14
Population: The Intent-to-Treat (RI/ST) analysis set included all the participants who received at least one dose of study medication in run-in phase or stabilization phase. "n" signifies those participants who were evaluated for this measure at the specified time point. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone: Run-in or Stabilization Phase: Paliperidone extended-release (ER) oral tablet was administered at a starting dose of 3 milligram (mg) once daily for 8 weeks. Dose was increased from 3 mg/day after 5 days based on Investigator's discretion, up to maximum of 12 mg/day.
Arm/Group | Paliperidone: Run-in or Stabilization Phase
Number analyzed (Participants) | 201
Units on a scale
  Baseline (n=201) | 89.5 (12.48)
  Change at Week 14 (n=200) | -30.8 (18.55)

3. Secondary Outcome: Double Blind (DB) Phase: Change From DB Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at DB Endpoint
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Change at DB endpoint was calculated as value at interim analysis data cut-off (09 November 2012) minus value at DB Baseline (Day 1 of week 15).
Time Frame: DB Baseline (Day 1 of Week 15) up to DB endpoint (study completion [09 November 2012] [Approximately 1 year])
Population: The Intent-to-Treat DB analysis set included all the participants who were randomized into the DB phase and who received at least one dose of DB study medication. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Units on a scale
  Baseline | 53.4 (9.71) [9. to NA] | 51.5 (9.50) [29.0 to 77.0]
  Change at DB endpoint | 2.0 (12.67) | 16.9 (16.16)

4. Secondary Outcome: Run-In and Stabilization Phase: Number of Participants Assessed With Categorical Scores Based on Clinical Global Impression-Severity Scale (CGI-S)
Description: The CGI-S is a 7-point clinician-rated scale to assess severity of participant's current illness state, ranging from (1)Normal, not ill at all, (2)Borderline mentally ill, (3)Mildly ill, (4)Moderately ill, (5)Markedly ill, (6)Severely ill, (7)Among the most severely ill.
Time Frame: Baseline and Week 14
Population: The Intent-to-Treat (RI/ST) analysis set included all the participants who received at least one dose of study medication in run-in phase or stabilization phase. "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Number; unit: Participants
Arm/Group | Paliperidone: Run-in or Stabilization Phase
Number analyzed (Participants) | 201
Participants
  Not ill: Baseline (n=201) | 0 (12.48)
  Not ill: Week 14 (n= 135) | 2 (18.49)
  Very Mild: Baseline (n= 201) | 0
  Very Mild: Week 14 (n= 135) | 37
  Mild: Baseline (n= 201) | 3
  Mild: Week 14 (n= 135) | 65
  Moderate: Baseline (n= 201) | 41
  Moderate: Week 14 (n= 135) | 27
  Marked: Baseline (n= 201) | 91
  Marked: Week 14 (n= 135) | 4
  Severe: Baseline (n= 201) | 66
  Severe: Week 14 (n= 135) | 0
  Extremely Severe: Baseline (n= 201) | 0
  Extremely Severe: Week 14 (n= 135) | 0

5. Secondary Outcome: Double Blind (DB) Phase: Change From DB Baseline in Clinical Global Impression-Severity Scale (CGI-S) Total Score at DB Endpoint
Description: CGI-S is a 7-point clinician-rated scale to assess severity of participant's current illness state, ranging from (1)Normal, not ill at all, (2)Borderline mentally ill, (3)Mildly ill, (4)Moderately ill, (5)Markedly ill, (6)Severely ill, (7)Among the most severely ill. Change at DB endpoint was calculated as value at interim analysis data cut-off (09 November 2012) minus value at DB Baseline (Day 1 of week 15).
Time Frame: DB Baseline (Day 1 of Week 15) up to DB endpoint (study completion [09 November 2012] [Approximately 1 year])
Population: The Intent-to-Treat DB analysis set included all the participants who were randomized into the DB phase and who received at least one dose of DB study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Units on a scale
  Baseline | 3.0 (0.88) [9. to NA] | 2.9 (0.70) [29.0 to 77.0]
  Change at DB endpoint | 0.1 (0.91) | 1.1 (1.11)

6. Secondary Outcome: Run-In and Stabilization Phase: Change From Baseline in Personal and Social Performance (PSP) Scale Total Score at Week 14
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty). Percentage of participants achieving improvement in PSP score by at least one category was reported.
Time Frame: Baseline and Week 14
Population: The Intent-to-Treat (RI/ST) analysis set included all the participants who received at least one dose of study medication in run-in phase or stabilization phase. "n" signifies those participants who were evaluated for this measure at the specified time point. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone: Run-in or Stabilization Phase
Number analyzed (Participants) | 201
Units on a scale
  Baseline (n=201) | 43.6 (13.96)
  Change at Week 14 (n=200) | 20.9 (17.55)

7. Secondary Outcome: Double Blind (DB) Phase: Change From DB Baseline in Personal and Social Performance (PSP) Scale Total Score at DB Endpoint
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty). Percentage of participants achieving improvement in PSP score by at least one category was reported. Change at DB endpoint was calculated as value at interim analysis data cut-off (09 November 2012) minus value at DB Baseline (Day 1 of week 15).
Time Frame: DB Baseline (Day 1 of Week 15) up to DB endpoint (study completion [09 November 2012] [Approximately 1 year])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Units on a scale
  Baseline | 69.3 (11.17) [9. to NA] | 69.9 (9.37) [29.0 to 77.0]
  Change at DB Endpoint | -2.9 (12.87) | -10.7 (14.99)

8. Secondary Outcome: Run-In and Stabilization Phase: Change From Baseline in Sleep Quality Based on Visual Analog Scale (VAS) at Week 14
Description: Sleep quality was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how well they slept in the previous 7 days (from 0: "very badly" to 100: "very well").
Time Frame: Baseline and Week 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone: Run-in or Stabilization Phase
Number analyzed (Participants) | 201
Millimeter (mm)
  Baseline (n=201) | 63.4 (24.60)
  Change at Week 14 (n=192) | 12.1 (29.13)

9. Secondary Outcome: Double Blind (DB) Phase: Change From DB Baseline in Sleep Quality Based on Visual Analog Scale (VAS) at DB Endpoint
Description: Sleep quality was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how well they slept in the previous 7 days (from 0: "very badly" to 100: "very well"). Change at DB endpoint was calculated as value at interim analysis data cut-off (09 November 2012) minus value at DB Baseline (Day 1 of week 15).
Time Frame: DB Baseline (Day 1 of Week 15) up to DB endpoint (study completion [09 November 2012] [Approximately 1 year])
Population: The Intent-to-Treat DB analysis set included all the participants who were randomized into the DB phase and who received at least one dose of DB study medication. "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Millimeter (mm)
  Baseline (n= 64, 71) | 77.5 (20.45) [9. to NA] | 81.9 (14.82) [29.0 to 77.0]
  Change at DB Endpoint (n= 60, 69) | -3.8 (20.02) | -22.4 (27.88)

10. Secondary Outcome: Run-In and Stabilization Phase: Change From Baseline in Daytime Drowsiness Based on Visual Analog Scale (VAS) at Week 14
Description: Daytime drowsiness was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how often they felt drowsy in the previous 7 days (from 0: "very badly" to 100: "very well").
Time Frame: Baseline and Week 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone: Run-in or Stabilization Phase
Number analyzed (Participants) | 201
Millimeter (mm)
  Baseline (n=201) | 32.8 (27.03)
  Change at Week 14 (n=192) | -7.3 (33.73)

11. Secondary Outcome: Double Blind (DB) Phase: Change From DB Baseline in Daytime Drowsiness Based on Visual Analog Scale (VAS) at DB Endpoint
Description: Daytime drowsiness was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how often they felt drowsy in the previous 7 days (from 0: "very badly" to 100: "very well"). Change at DB endpoint was calculated as value at interim analysis data cut-off (09 November 2012) minus value at DB Baseline (Day 1 of week 15).
Time Frame: DB Baseline (Day 1 of Week 15) up to DB endpoint (study completion [09 November 2012] [Approximately 1 year])
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Millimeter (mm)
  Baseline (n= 64, 71) | 22.9 (24.24) [9. to NA] | 24.4 (22.93) [29.0 to 77.0]
  Change at DB Endpoint (n= 60, 69) | 3.1 (23.18) | 1.2 (28.50)

12. Secondary Outcome: Double Blind (DB) Phase: Median Time to Relapse (Final Analysis)
Description: A relapse is defined as any one of the following: 1. involuntary or voluntary psychiatric hospitalization 2. deliberate self-injury or violent behavior; 3. Suicidal or homicidal ideation and clinically significant aggressive behavior; 4. 25 percent (%) increase in Positive and Negative Syndrome Scale (PANSS) total score for 2 consecutive assessments for participants whose score was greater than 40 at randomization, or a 10-point increase for participants who scored less than or equal to (≤) 40 at randomization; 5. increase for 2 consecutive assessments in PANSS items (delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, hostility or uncooperativeness) to greater than or equal to (≥) 5 for participants who scored ≤3 at randomization, or to ≥6 for participants with initial score of 4. Independent Data Monitoring Committee performed final analysis at the end of double-blind treatment (09 November 2012).
Time Frame: DB Baseline (Day 1 of Week 15) up to study completion (09 November 2012) (Approximately 1 year)
Population: The Intent-to-Treat DB analysis set included all the participants who were randomized into the DB phase and who received at least one dose of DB study medication up to final analysis cut-off date (09-Nov-2012).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase
Number analyzed (Participants) | 64 | 71
Days | NA [NA to NA] — Median time was not reached as data was not matured at the time of the analysis, hence no data could be reported. | 52.0 [29.0 to 77.0]

13. Secondary Outcome: Open-label Extension (OLE) Phase: Change From OLE Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at OLE Endpoint
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Change at OLE endpoint was calculated as value at OLE endpoint (24 weeks after DB phase (26 April 2013) minus value at OLE Baseline (09 November 2012).
Time Frame: OLE Baseline (09 November 2012) up to OLE endpoint (that is, up to 24 Weeks [26 April 2013] from DB endpoint)
Population: The Intent-to-Treat (ITT) OLE analysis set included all participants who received at least one dose of OLE medication as recorded on the electronic case report form (eCRF). LOCF method was used to impute missing values. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Number analyzed (Participants) | 46 | 59
Units on a scale
  Baseline | 56.5 (14.86) [9. to NA] | 67.2 (14.67) [29.0 to 77.0]
  Change at OLE endpoint | -3.9 (11.30) | -15.4 (12.41)

14. Secondary Outcome: Open-label Extension (OLE) Phase: Change From OLE Baseline in Clinical Global Impression-Severity Scale (CGI-S) Total Score at OLE Endpoint
Description: CGI-S is a 7-point clinician-rated scale to assess severity of participant's current illness state, ranging from (1)Normal, not ill at all, (2)Borderline mentally ill, (3)Mildly ill, (4)Moderately ill, (5)Markedly ill, (6)Severely ill, (7)Among the most severely ill. Change at OLE endpoint was calculated as value at OLE endpoint (24 weeks after DB phase (26 April 2013) minus value at OLE Baseline (09 November 2012).
Time Frame: OLE Baseline (09 November 2012) up to OLE endpoint (that is, up to 24 Weeks [26 April 2013] from DB endpoint)
Population: The ITT OLE analysis set included all participants who received at least one dose of OLE medication as recorded on the electronic case report form (eCRF). LOCF method was used to impute missing values. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Number analyzed (Participants) | 46 | 59
Units on a scale
  Baseline | 3.1 (1.02) [9. to NA] | 3.9 (0.98) [29.0 to 77.0]
  Change at OLE endpoint | -0.2 (0.78) | -0.9 (0.97)

15. Secondary Outcome: Open-label Extension (OLE) Phase: Change From OLE Baseline in Personal and Social Performance (PSP) Scale Total Score at OLE Endpoint
Description: The PSP is 100-point validated clinician-rated scale that assesses degree of difficulty in 4 areas of functioning: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors rated on 6-point scale (1=absent to 6=very severe).Total transformed score from 1 to 100 is generated from raw score based on clinical interpretation of scores generated in 4 areas of functioning, with higher transformed score indicating better function. Total score is divided into 3 levels: 71-100 (mild difficulty); 31-70 (marked difficulty) and 1-30 (severe difficulty). Percentage of participants achieving improvement in PSP score by at least one category was reported. Change at OLE endpoint was calculated as value at OLE endpoint (24 weeks after DB phase (26 April 2013) minus value at OLE Baseline (09 November 2012).
Time Frame: OLE Baseline (09 November 2012) up to OLE endpoint (that is, up to 24 Weeks [26 April 2013] from DB endpoint)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Number analyzed (Participants) | 46 | 59
Units on a scale
  Baseline | 66.8 (15.68) [9. to NA] | 60.6 (15.63) [29.0 to 77.0]
  Change at OLE endpoint | 10.88 (3.1) | 10.7 (14.01)

ADVERSE EVENTS:
Description: Safety analysis set included all the participants who were randomized into the double-blind phase and received at least 1 dose of double-blind medication.
Arm/Group | Paliperidone: Run-in or Stabilization Phase | Paliperidone: Double Blind (DB) Phase | Placebo: DB Phase | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase | Placebo DB/Paliperidone OL Extension Phase
Serious Adverse Events (participants affected / at risk) | 2/201 | 2/64 | 8/71 | 2/47 | 0/59
Other Adverse Events (participants affected / at risk) | 141/201 | 12/64 | 12/71 | 6/47 | 14/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone: Run-in or Stabilization Phase (N=201) | Paliperidone: Double Blind (DB) Phase (N=64) | Placebo: DB Phase (N=71) | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase (N=47) | Placebo DB/Paliperidone OL Extension Phase (N=59)
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Hallucination, Auditory (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 1 | 5 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone: Run-in or Stabilization Phase (N=201) | Paliperidone: Double Blind (DB) Phase (N=64) | Placebo: DB Phase (N=71) | Paliperidone DB/Paliperidone Open-label (OL) Extension Phase (N=47) | Placebo DB/Paliperidone OL Extension Phase (N=59)
Tachycardia (Cardiac disorders) | 12 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 19 | 1 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 13 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 19 | 1 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 12 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 17 | 0 | 2 | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 1 | 1 | 1 | 1
Weight Increased (Investigations) | 13 | 1 | 1 | 0 | 2
Akathisia (Nervous system disorders) | 52 | 3 | 0 | 1 | 3
Dyskinesia (Nervous system disorders) | 11 | 0 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 11 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 11 | 1 | 0 | 1 | 1
Hypertonia (Nervous system disorders) | 14 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 19 | 0 | 0 | 1 | 3
Tremor (Nervous system disorders) | 24 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 21 | 1 | 6 | 1 | 1
Restlessness (Psychiatric disorders) | 12 | 1 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Independent Data Monitoring Committee (IDMC) conducted an interim analysis after 61st relapse in double-blind (DB) phase and DB phase completed on 09-Nov-2012 based on positive results of interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wishes to publish information from study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. If requested by the Sponsor, investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application. Investigators will not publish data derived from individual site until Sponsor confirms there will be no multi-center study publication.